CLINICAL TRIAL: NCT05042791
Title: SRT Versus WBRT Combined With Pyrrotinib and Capecitabine in the Treatment of HER2-positive Advanced Breast Cancer Patients With Brain Metastases: A Randomized Controlled, Prospective Clinical Study
Brief Title: A Study of Pyrotinib Plus Capecitabine Combined With SRT in HER2+ MBC With Brain Metastases
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangxi Provincial Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20210901-jiangchunling
Record Dates: First submitted 2021-09-06; First posted 2021-09-13 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: HER2-positive Metastatic Breast Cancer
MeSH Terms: interventions — pyrotinib; Capecitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SRT combined with pyrotinib and capecitabine (Experimental): SRT: SRT needs to be comprehensively considered based on the size, number, and location of the lesion, and SRS and FSRT are performed according to clinical needs.
  Pyrotinib:400mg/d,q.d.,p.o. A course of treatment need 21days. Capecitabine:1000mg/m2,bid,from day1-day14, A course of treatment need 21 days.
  Interventions: Combination Product: radiation combined with pyrotinib and capecitabine
- WBRT combined with pyrotinib and capecitabine (Active Comparator): WBRT: WBRT need to be considered based on the size, number, and location of the lesion.
  Pyrotinib:400mg/d,q.d.,p.o. A course of treatment need 21days. Capecitabine:1000mg/m2,bid,from day1-day14, A course of treatment need 21 days.
  Interventions: Combination Product: radiation combined with pyrotinib and capecitabine

INTERVENTIONS:
Combination Product: radiation combined with pyrotinib and capecitabine — This study selects different radiation (SRT or WBRT) combined with pyrotinib and capecitabine to treat HER2-positive advanced breast cancer patients with brain metastases

SUMMARY:
This study evaluates the efficacy and safety of SRT combined with pyrotinib and capecitabine in the treatment of patients with HER2-positive advanced breast cancer patients with brain metastases.

DETAILED DESCRIPTION:
Brain metastases occur in 30-50% of patients with metastatic HER2-positive breast cancer. In the case of multiple brain metastases, radiation therapy is the preferred therapeutic approaches. However, the side effects of WBRT for long-lived patients are also obvious, such as irreversible decline in cognitive function and decline in memory function. WBRT can also cause extensive hair loss and extensive white matter lesions on imaging. Pyrotinib as an oral tyrosine kinase inhibitor has good efficacy and safety in patients with breast cancer brain metastases. Therefore, in order to reduce the impact of WBRT on the cognitive function, a phase II clinical study of SRT versus WBRT combined with pyrotinib and capecitabine in the treatment of MBC with brain metastases was carried out to explore the efficacy and safety of radiotherapy de-escalation therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age> 18 years old, female
2. KPS≥70
3. HER2-positive breast cancer is confirmed by the pathology laboratory with an immunohistochemical (IHC) score of 3+ and/or 2+ and a positive in situ hybridization (ISH) test (ISH amplification rate ≥ 2.0)
4. Brain metastasis confirmed by MRI, in line with the indications for whole brain radiotherapy
5. At least one measurable brain lesion exists according to the RECIST 1.1 standard
6. Unlimited number of previous chemotherapy lines
7. Have not used capecitabine in the past, or progressed 6 months after capecitabine stopped, or progressed after capecitabine as adjuvant therapy stopped for one year
8. The expected survival period is more than 12 weeks
9. Patients must have adequate organ function, criteria as follows.

   1. Blood routine examination：Absolute Neutrophil Count (ANC)≥1.5×109/L；PLT ≥100×109/L； Hb ≥90g/L
   2. Blood chemistry test：TBIL ≤1.5 times the upper limit of normal (ULN); ALT and AST≤3 times ULN; For patients with liver metastases, ALT and AST≤5×ULN; BUN and Cr≤1×ULN and creatinine clearance ≥50mL/min (CockcroftGault formula);
   3. Ultrasonic cardiogram: LVEF≥50%
   4. 12-lead ECG: The QT interval (QTcF) corrected by Fridericia's method is < 470 ms
10. Patients with known hormone receptor status
11. Patients need to voluntarily join this study after they fully understand and sign the informed consent form. Patients need to have good compliance and be willing to cooperate with follow-up.

Exclusion Criteria:

1. Patients with brain metastases with extensive meningeal metastasis
2. Brain metastases within 5 mm of the hippocampus
3. There are many factors that affect the administration and absorption of drugs, for example: inability to swallow, chronic diarrhea and intestinal obstruction
4. Those who have received chemotherapy, surgical treatment (excluding local puncture) or molecular targeted therapy within 4 weeks before enrollment; those who have received anti-tumor endocrine therapy after the screening period
5. Participated in other drug clinical trials within 4 weeks before enrollment
6. Have used or are currently using HER2 tyrosine kinase inhibitors (lapatinib, niratinib, pyrotinib, etc.)
7. Suffered from other malignant tumors in the past 5 years, excluding cured cervical carcinoma in situ, skin basal cell carcinoma or skin squamous cell carcinoma
8. Receive any other anti-tumor therapy at the same time
9. Those who are known to have a history of allergies to the drug; have a history of immunodeficiency, including positive HIV tests, HCV, active hepatitis B, or other acquired or congenital immunodeficiency diseases, or organ transplants history
10. Have ever suffered from any heart disease, including: (1) arrhythmia requiring medication or clinical significance; (2) myocardial infarction; (3) heart failure; (4) anyone judged by the researcher as unsuitable for participation becase of other heart diseases in this trial, etc.
11. Female patients during pregnancy and lactation, female patients with fertility and a positive baseline pregnancy test, or female patients of childbearing age who are unwilling to take effective contraceptive measures during the entire trial period
12. According to the judgment of the investigator, there are accompanying diseases that seriously endanger the safety of the patient or affect the completion of the study (including but not limited to severe hypertension that cannot be controlled by drugs, severe diabetes, active infection, etc.)
13. The patient has not recovered from the toxicity of the previous treatment to grade 0-1 (except for hair loss)
14. Have a clear history of neurological or psychiatric disorders, including epilepsy or dementia
15. Concomitant use of CYP3A4 inhibitors or inducers or drugs that prolong the QT interval
16. Any other circumstances that are not suitable for inclusion in this study (investigator assessment)

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 362 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
CNS-ORR | Estimated up to 1 year
  Objective response rate of central nervous system

CONTACTS AND LOCATIONS:
Overall Officials: Chunling Jiang, Principal Investigator — Jiangxi Provincial Cancer Hospital
Locations (1):
- Jiangxi Cancer Hospital of Nanchang University, Nanchang, Jiangxi, China

REFERENCES:
- [Derived] Dai L, Gao T, Guo R, Chen Y, Wang J, Zhou S, Tang Y, Chen D, Huang S. Efficacy and safety of pyrotinib-based regimens in HER2 positive metastatic breast cancer: A retrospective real-world data study. Neoplasia. 2024 Oct;56:101029. doi: 10.1016/j.neo.2024.101029. Epub 2024 Jul 17. PMID 39024777